CLINICAL TRIAL: NCT01284634
Title: A Randomised, Partially-blind, Placebo-controlled, Pilot, Dose-ranging Study To Assess The Effect Of Cannabidiol (CBD) On Liver Fat Levels In Subjects With Fatty Liver Disease.
Brief Title: Study to Evaluate the Effect of GWP42003 on Liver Fat Levels in Participants With Fatty Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GW Research Ltd (Industry)
Responsible Party: Sponsor
Organization: GWResearch (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWMD09112; 2009-017080-41 (EudraCT Number)
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Results first posted 2014-01-20 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Fatty Liver
Keywords: Cannabidiol; Fatty liver; Diabetes; Body fat
MeSH Terms: conditions — Fatty Liver; Diabetes Mellitus | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study was partially-blinded. Due to the varying numbers of capsules administered, participants and investigators were not blinded to the treatment cohort (one, two or four capsules), but were blinded to the treatment allocation within each cohort (GWP42003 or placebo)
Oversight: Data Monitoring Committee: No

ARMS (4):
- GWP42003 200 milligrams (mg)/day Dose (Experimental): Participants self-administered one x 100 mg GWP42003 capsule twice daily for 8 weeks (the first dose was 30 minutes before breakfast [fasted] and the second was 30 minutes before the evening meal [typically 12 hours apart]).
  Interventions: Drug: GWP42003 200 mg/day Dose
- GWP42003 400 mg/day Dose (Experimental): Participants self-administered two x 100 mg GWP42003 capsules twice daily for 8 weeks (the first dose was 30 minutes before breakfast [fasted] and the second was 30 minutes before the evening meal [typically 12 hours apart]).
  Interventions: Drug: GWP42003 400 mg/day Dose
- GWP42003 800 mg/day Dose (Experimental): Participants self-administered four x 100 mg GWP42003 capsules twice daily for 8 weeks (the first dose was 30 minutes before breakfast [fasted] and the second was 30 minutes before the evening meal [typically 12 hours apart]).
  Interventions: Drug: GWP42003 800 mg/day Dose
- Placebo (Experimental): Participants self-administered one, two or four placebo capsules twice daily, for 8 weeks (the first dose was 30 minutes before breakfast [fasted] and the second was 30 minutes before the evening meal [typically 12 hours apart]). Each capsule exactly matched the GWP42003 capsules in terms of appearance, size, smell and taste.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GWP42003 200 mg/day Dose — GWP42003 was presented as Licaps® size double zero (Size 00) hard gelatin capsules containing 100 mg of CBD dissolved in vehicle (Gelucire 44/14).
  Other Names: Cannabidiol, CBD
  Arms: GWP42003 200 milligrams (mg)/day Dose
Drug: GWP42003 400 mg/day Dose — GWP42003 was presented as Licaps® Size 00 hard gelatin capsules containing 100 mg of CBD dissolved in vehicle (Gelucire 44/14).
  Other Names: Cannabidiol, CBD
  Arms: GWP42003 400 mg/day Dose
Drug: GWP42003 800 mg/day Dose — GWP42003 was presented as Licaps® Size 00 hard gelatin capsules containing 100 mg of CBD dissolved in vehicle (Gelucire 44/14).
  Other Names: Cannabidiol, CBD
  Arms: GWP42003 800 mg/day Dose
Drug: Placebo — Placebo was presented as Licaps® Size 00 hard gelatin capsules containing excipients (Gelucire 44/14).
  Other Names: Placebo control
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of GWP42003 on liver triglyceride (liver fat) in participants with fatty liver disease (FLD).

DETAILED DESCRIPTION:
This study was conducted as a 10-week (eight-week treatment period and one-week safety follow-up), randomized, partially-blind study that evaluated the effect of GWP42003 in participants with raised liver triglycerides (liver fat ≥5%). Participants were clinically diagnosed with FLD and had liver fat levels ≥5% as measured by Magnetic Resonance Imaging/ Magnetic Resonance Scanning (MRI/MRS), or were willing to undergo MRI/MRS scan at the screening visit to confirm a liver fat content of ≥5%. Eligible participants entered the study at a screening visit (Day -10 to -2) and then returned for a fasted baseline visit (Day 1), a mid-treatment visit (Day 29) and an end of treatment visit (Day 57). Safety follow-up telephone calls took place throughout the treatment period up to Day 64 after completion of treatment or seven days after date of last dose/withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Participant gave informed consent for participation in the study.
* Participant was aged 18 years or above.
* Participant had documented evidence of liver fat content ≥5% as measured by MRI/MRS scanning or a biopsy within two months prior to screening, or willing to undergo an MRI/MRS scan at Visit 1 (Day -10 to -2) to confirm a liver fat content of ≥5%.
* Participant had, in the opinion of the investigator, no changes in levels of exercise or diet for four weeks (as assessed by the physical activity questionnaire and food frequency questionnaire) prior to the start of treatment, and participant agreed to keep stable for the duration of the study.
* Participant was able (in the investigator's opinion) and willing to comply with all study requirements.
* Participant was willing for his or her name to be notified to the responsible authorities for participation in this study, as applicable.
* Participant was willing to allow his or her primary care practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* Participant had clinical diagnosis or treatment for Type I/II diabetes.
* Participant had received an unapproved investigational medicinal product (IMP) within the 30 days prior to the screening visit.
* Participant was receiving a prohibited medication and unwilling to stop for 14 days prior to the screening visit and for the duration of the study.
* Participant was using or had used recreational cannabis, medicinal cannabis, or cannabinoid medications (including Sativex) within one month prior to study entry and unwilling to abstain for the duration of the study.
* Participant had any known or suspected history of alcohol or substance abuse, or epilepsy or recurrent seizures.
* Participant had any known or suspected history of major depression sufficient to require treatment or disrupt ordinary life (excluding episodes of reactive depression, in the opinion of the investigator).
* Participant had clinically significant cardiac, renal, or hepatic impairment, in the opinion of the investigator.
* Participant had known history of Hepatitis B or C.
* Participant had genetic dyslipidaemia, in the opinion of the Investigator.
* Participant had any other significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, influence the result of the study, or affect the participant's ability to participate in the study.
* Participant had any known or suspected hypersensitivity to cannabinoids or any of the excipients of the IMP(s).
* Participant had presence of any metal implants.
* Participant had any known or suspected history of claustrophobia.
* Female participants of child bearing potential not able or willing to use effective contraception for the duration of the study and for three months thereafter, or male participants whose partner was of child bearing potential, who was not willing to ensure that they or their partner would use effective contraception during the study and for three months thereafter.
* Female participant who was pregnant, lactating or planning pregnancy during the course of the study and for three months thereafter.
* Participants who weighed >150 kilograms (kg).
* Participant had any abnormalities following a physical examination that, in the opinion of the investigator, prevented the participant from safe participation in the study.
* Participant was unwilling to abstain from donation of blood during the study.
* Participant had planned travel outside the country of residence during the study.
* Participant had previously enrolled into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-05-03 (Actual); Primary Completion 2012-07-13 (Actual); Study Completion 2012-07-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - London
  - Manchester

RESULTS

PARTICIPANT FLOW:
Groups:
- GWP42003 200 Milligram (mg)/Day Dose: Participants self-administered one 100 mg GWP42003 capsule twice daily for 8 weeks (the first dose was 30 minutes before breakfast [fasted] and the second was 30 minutes before the evening meal [typically 12 hours apart]).
- Placebo: Participants self-administered one, two or four placebo capsules twice daily, for 8 weeks (the first dose was 30 minutes before breakfast [fasted] and the second was 30 minutes before the evening meal [typically 12 hours apart]).
Period: Overall Study
Arm/Group | GWP42003 200 Milligram (mg)/Day Dose | GWP42003 400 mg/Day Dose | GWP42003 800 mg/Day Dose | Placebo
Started | 7 | 6 | 7 | 5
Received at Least 1 Dose of Study Drug (Safety analysis set; analyzed as per actual treatment received.) | 7 | 6 | 7 | 5
Intent to Treat (ITT) Analysis Set (Randomized and received at least one dose of study medication and had on-treatment efficacy data.) | 7 | 6 | 7 | 5
Completed | 6 | 6 | 5 | 4
Not Completed | 1 | 0 | 2 | 1
Not completed — Adverse Event | 1 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: Participants who received at least 1 dose of investigational medicinal product (IMP); analyzed as per actual treatment received.
Groups:
- GWP42003 200 mg/Day Dose: Participants self-administered one 100 mg GWP42003 capsule twice daily for 8 weeks (the first dose was 30 minutes before breakfast [fasted] and the second was 30 minutes before the evening meal [typically 12 hours apart]).
- Total: Total of all reporting groups
Arm/Group | GWP42003 200 mg/Day Dose | GWP42003 400 mg/Day Dose | GWP42003 800 mg/Day Dose | Placebo | Total
Number analyzed (Participants) | 7 | 6 | 7 | 5 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.69 (14.62) | 49.08 (7.72) | 46.90 (12.57) | 50.41 (18.41) | 46.39 (13.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 2 | 4 | 13
  Male | 2 | 4 | 5 | 1 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline To The End Of Treatment (EOT) In Mean Liver Triglyceride Levels
Description: Liver triglyceride levels were measured by Magnetic Resonance Imaging/Magnetic Resonance Scanning and the percent change from baseline to EOT in group mean levels was investigated. A reduction from baseline, that is, a negative value, indicates an improvement in condition.
Time Frame: Baseline to EOT (Day 57) or Early Termination (ET)
Population: ITT analysis set: All participants who were randomized, received at least one dose of study medication, and had on-treatment efficacy data. Participants who did not have any relevant post-randomization efficacy data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | GWP42003 200 mg/Day Dose | GWP42003 400 mg/Day Dose | GWP42003 800 mg/Day Dose | Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 5
percentage change | -0.68 (4.97) | -0.28 (8.60) | 0.65 (5.28) | 6.36 (17.97)
Statistical Analysis 1: Comparison: GWP42003 200 mg/Day Dose vs Placebo; The EOT liver triglyceride levels were analyzed using a linear regression model, with EOT liver triglyceride levels as the dependent variable, dose of GWP42003 as regressor, baseline liver triglyceride levels as a covariate, and gender as a factor; Test type: Superiority or Other; p = 0.222, Regression, Linear; Mean Difference (Final Values) = -6.89, 90% CI 2-sided [-16.35 to 2.56], Standard Error of Mean 5.454
Statistical Analysis 2: Comparison: GWP42003 400 mg/Day Dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.133, Regression, Linear; Mean Difference (Final Values) = -9.35, 90% CI 2-sided [-19.66 to 0.95], Standard Error of Mean 5.943
Statistical Analysis 3: Comparison: GWP42003 800 mg/Day Dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.302, Regression, Linear; Mean Difference (Final Values) = -6.54, 90% CI 2-sided [-17.22 to 4.14], Standard Error of Mean 6.158

2. Secondary Outcome: Change From Baseline To The EOT In Mean Serum Total Cholesterol Levels
Description: A fasting blood sample was taken for the measurement of serum total cholesterol. A reduction from baseline, that is, a negative value, indicates an improvement in condition.
Time Frame: Baseline to EOT (Day 57) or ET
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimole (mmol)/l
Arm/Group | GWP42003 200 mg/Day Dose | GWP42003 400 mg/Day Dose | GWP42003 800 mg/Day Dose | Placebo
Number analyzed (Participants) | 7 | 6 | 7 | 5
millimole (mmol)/l | 0.07 (0.76) | 0.03 (0.51) | -0.14 (0.31) | -0.62 (1.00)

3. Secondary Outcome: Change From Baseline To The EOT In Mean Serum High Density Lipoprotein (HDL)-Cholesterol(C) Levels
Description: A fasting blood sample was obtained for the measurement of HDL-C. An increase from baseline, that is, a positive value, indicates an improvement in condition.
Time Frame: Baseline to EOT (Day 57) or ET
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | GWP42003 200 mg/Day Dose | GWP42003 400 mg/Day Dose | GWP42003 800 mg/Day Dose | Placebo
Number analyzed (Participants) | 7 | 6 | 7 | 5
mmol/l | 0.07 (0.15) | 0.08 (0.15) | 0.06 (0.17) | -0.14 (0.23)

4. Secondary Outcome: Change From Baseline To The EOT In Mean Serum Low-Density Lipoprotein (LDL)-C Levels
Description: A fasting blood sample was obtained for the measurement of LDL-C. An increase from baseline, that is, a positive value, indicates an improvement in condition.
Time Frame: Baseline to EOT (Day 57) or ET
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | GWP42003 200 mg/Day Dose | GWP42003 400 mg/Day Dose | GWP42003 800 mg/Day Dose | Placebo
Number analyzed (Participants) | 7 | 6 | 7 | 5
mmol/l | 0.11 (0.631) | 0.08 (0.407) | 0.00 (0.432) | -0.34 (0.737)

5. Secondary Outcome: Change From Baseline To The EOT In Mean Serum HDL: Low Density Lipoprotein (LDL)-Cholesterol (C) Ratio
Description: A fasting blood sample was obtained for the measurement of HDL-C and LDL-C, allowing the HDL:LDL cholesterol ratio to be calculated. An increase from baseline, that is, a positive value, indicates an improvement in condition.
Time Frame: Baseline to EOT (Day 57) or ET
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change in ratio
Arm/Group | GWP42003 200 mg/Day Dose | GWP42003 400 mg/Day Dose | GWP42003 800 mg/Day Dose | Placebo
Number analyzed (Participants) | 7 | 6 | 7 | 5
change in ratio | -0.02 (0.13) | -0.00 (0.08) | 0.03 (0.09) | 0.01 (0.06)

6. Secondary Outcome: Change From Baseline To The EOT In Mean Serum Triglyceride Levels
Description: A fasting blood sample was obtained for the measurement of serum triglycerides. A reduction from baseline, that is, a negative value, indicates an improvement in condition.
Time Frame: Baseline to EOT (Day 57) or ET
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | GWP42003 200 mg/Day Dose | GWP42003 400 mg/Day Dose | GWP42003 800 mg/Day Dose | Placebo
Number analyzed (Participants) | 7 | 6 | 7 | 5
mmol/l | -0.40 (1.05) | -0.29 (0.82) | -0.50 (1.16) | -0.28 (0.39)

ADVERSE EVENTS:
Time Frame: Day 1 through Day 77
Description: Safety analysis set: All randomized participants who received at least one dose of IMP were included and analyzed according to the treatment received.
Groups:
- GWP42003 200 mg/Day Dose: Participants self-administered one x 100 mg GWP42003 capsule twice daily for 8 weeks (the first dose was 30 minutes before breakfast [fasted] and the second was 30 minutes before the evening meal [typically 12 hours apart]).
- 800 mg GWP42003: Participants self-administered four x 100 mg GWP42003 capsules twice daily for 8 weeks (the first dose was 30 minutes before breakfast [fasted] and the second was 30 minutes before the evening meal [typically 12 hours apart]).
Arm/Group | GWP42003 200 mg/Day Dose | GWP42003 400 mg/Day Dose | 800 mg GWP42003 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 6/7 | 5/6 | 7/7 | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003 200 mg/Day Dose (N=7) | GWP42003 400 mg/Day Dose (N=6) | 800 mg GWP42003 (N=7) | Placebo (N=5)
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 5 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal hypermotility (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0
Product size issue (General disorders) | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0
Heart sounds abnormal (Investigations) | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 3 | 2 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1
Poor quality sleep (Nervous system disorders) | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.